CLINICAL TRIAL: NCT00000149
Title: Collaborative Initial Glaucoma Treatment Study (CIGTS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-50
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-06

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Adrenergic beta-Antagonists; Trabeculectomy

INTERVENTIONS:
Drug: Beta Blocker
Procedure: Trabeculectomy
Procedure: Argon Laser Trabeculoplasty

SUMMARY:
To compare the long-term effect of treating newly diagnosed open-angle glaucoma with standard medical treatment versus filtration surgery.

DETAILED DESCRIPTION:
Recent studies have challenged the conventional wisdom of treating all newly diagnosed open-angle glaucoma (OAG) with eyedrops; rather, these studies suggest that more effective control of glaucomatous damage can be obtained by immediate filtration surgery. In addition, increased attention to the impact of therapy on health-related quality of life has added another consideration in deciding upon appropriate treatment of such patients.

The Collaborative Initial Glaucoma Treatment Study (CIGTS), a randomized, controlled clinical trial, is being conducted to determine whether patients with newly diagnosed OAG are best managed by the conventional approach of topical pharmacologic agents or by immediate filtration surgery. Eligible patients were randomized to receive either a stepped medication treatment regimen or filtration surgery to control their OAG. Sample size requirements indicated that 300 patients were needed for each treatment approach; a total of 607 patients were ultimately recruited for the CIGTS.

Patients randomized to the medication treatment arm are receiving a stepped regimen of topical medications, beginning with a single agent (typically a beta blocker), with additional medications added upon documented lack of intraocular pressure control or evidence of progressive visual field loss. If medications fail to control the patient's OAG, a series of treatment steps begin with argon laser trabeculoplasty and conclude with trabeculectomy.

In the surgical treatment arm, patients underwent immediate trabeculectomy and, with documented failure, proceed to argon laser trabeculectomy, then conclude with medications. Patients, rather than eyes, are randomized to the two treatment arms; if both eyes are eligible for treatment, the treatment course for both eyes is the same and was determined in the randomization.

Following randomization, participating community ophthalmologists affiliated with the study have been allowed to manage the medical and surgical care of study patients. However, all patients are seen at the Clinical Centers for standardized followup examinations at 3 and 6 months after treatment and every 6 months thereafter; in addition, patients randomized to the surgical arm will receive, at a minimum, postsurgical followup at 1 day, 1 week, and 1 month. At the Clinical Center visits, examination of the eye(s) includes evaluation of visual acuity, visual field, and intraocular pressure. The results of these tests determine whether treatment should be changed. In addition, before and at regular intervals after treatment, patients are being interviewed by telephone to assess their health-related quality of life. A questionnaire that includes the Sickness Impact Profile, Visual Activities Questionnaire, and other components is being used.

ELIGIBILITY:
Patients must be at least 25 years old with an intraocular pressure of 20 mm Hg or greater and evidence of optic nerve damage and/or visual field loss in one or both eyes. The ocular findings must exclude causes of glaucoma other than primary open-angle glaucoma, pigmentary glaucoma, or pseudoexfoliation glaucoma.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-10

REFERENCES:
- [Background] Janz N; Wren PA; CIGTS Study Group; Implementing quality of life in a clinical trial, in Anderson DR, Drance SM (eds)., The Collaborative Initial Glaucoma Treatment Study. Encounters in Glaucoma Research 3: How to Ascertain Progression and Outcome, 1996:45-62
- [Background] Lichter PR; Mills RP; CIGTS Study Group; Quality of life study - determination of progression, in Anderson DR, Drance SM (eds)., Encounters in Glaucoma Research 3: How to Ascertain Progression and Outcome, Amsterdam, Kugler Publications, 1996:149-163
- [Background] Mills RP, Janz NK, Wren PA, Guire KE. Correlation of visual field with quality-of-life measures at diagnosis in the Collaborative Initial Glaucoma Treatment Study (CIGTS). J Glaucoma. 2001 Jun;10(3):192-8. doi: 10.1097/00061198-200106000-00008. PMID 11442181
- [Background] Lichter PR, Musch DC, Gillespie BW, Guire KE, Janz NK, Wren PA, Mills RP; CIGTS Study Group. Interim clinical outcomes in the Collaborative Initial Glaucoma Treatment Study comparing initial treatment randomized to medications or surgery. Ophthalmology. 2001 Nov;108(11):1943-53. doi: 10.1016/s0161-6420(01)00873-9. PMID 11713061
- [Background] Janz NK, Wren PA, Lichter PR, Musch DC, Gillespie BW, Guire KE, Mills RP; CIGTS Study Group. The Collaborative Initial Glaucoma Treatment Study: interim quality of life findings after initial medical or surgical treatment of glaucoma. Ophthalmology. 2001 Nov;108(11):1954-65. doi: 10.1016/s0161-6420(01)00874-0. PMID 11713062
- [Background] Janz NK, Wren PA, Lichter PR, Musch DC, Gillespie BW, Guire KE. Quality of life in newly diagnosed glaucoma patients : The Collaborative Initial Glaucoma Treatment Study. Ophthalmology. 2001 May;108(5):887-97; discussion 898. doi: 10.1016/s0161-6420(00)00624-2. PMID 11320018
- [Background] Musch DC, Lichter PR, Guire KE, Standardi CL. The Collaborative Initial Glaucoma Treatment Study: study design, methods, and baseline characteristics of enrolled patients. Ophthalmology. 1999 Apr;106(4):653-62. doi: 10.1016/s0161-6420(99)90147-1. PMID 10201583
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114
- [Derived] Musch DC, Niziol LM, Gillespie BW, Lichter PR, Janz NK. Binocular Measures of Visual Acuity and Visual Field versus Binocular Approximations. Ophthalmology. 2017 Jul;124(7):1031-1038. doi: 10.1016/j.ophtha.2017.02.013. Epub 2017 Apr 10. PMID 28408039
- [Derived] Gillespie BW, Musch DC, Niziol LM, Janz NK. Estimating minimally important differences for two vision-specific quality of life measures. Invest Ophthalmol Vis Sci. 2014 Jun 6;55(7):4206-12. doi: 10.1167/iovs.13-13683. PMID 24906863
- [Derived] Musch DC, Gillespie BW, Palmberg PF, Spaeth G, Niziol LM, Lichter PR. Visual field improvement in the collaborative initial glaucoma treatment study. Am J Ophthalmol. 2014 Jul;158(1):96-104.e2. doi: 10.1016/j.ajo.2014.04.003. Epub 2014 Apr 12. PMID 24727262
- [Derived] Parrish RK 2nd, Feuer WJ, Schiffman JC, Lichter PR, Musch DC; CIGTS Optic Disc Study Group. Five-year follow-up optic disc findings of the Collaborative Initial Glaucoma Treatment Study. Am J Ophthalmol. 2009 Apr;147(4):717-724.e1. doi: 10.1016/j.ajo.2008.10.007. Epub 2009 Jan 18. PMID 19152871